CLINICAL TRIAL: NCT00584467
Title: Genetic and Inflammatory Markers in Cardiovascular Disease (GEM) Registry
Acronym: GEM
Status: Terminated | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 200513134
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Atherosclerosis
Keywords: GEM; Arteriosclerosis; biomarkers; Atherosclerosis
MeSH Terms: conditions — Atherosclerosis; Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood/serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an investigator initiated registry aimed at assembling a blood/serum and genomic resource (bank) of human blood samples with accompanying clinical data mainly from patients who are scheduled to undergo cardiac catheterization at UC Davis Medical Center, but may also include other eligible individuals. Funding is from institutional/divisional research funds.

DETAILED DESCRIPTION:
This study is aimed at assembling a blood/serum and genomic resource (bank) of human samples with accompanying clinical data mainly from patients who are scheduled to undergo cardiac catheterization at UC Davis Medical Center, but may also include other eligible individuals. These samples will be analyzed at UC Davis Medical Center for determination of biomarker levels, and concomitantly analyzed at UC San Francisco in an IRB-approved protocol at that institution for genetic analysis (UCSF IRB approval # for this study is H711-15138-03; protocol name is "Discovery of Gene Mutations and Polymorphisms that Contribute to the Risk of Atherosclerosis"; principal investigator is John P. Kane, MD). All samples sent to UCSF will be de-identified and catalogued using an alphanumeric code. A number of candidate genes will be studied to detect mutations and polymorphisms that could contribute to the risk of atherosclerosis. The technique of hybridization sequencing will be employed for this. The techniques of classical statistical genetics will be employed for both cosegregation analysis and for the genome search approach. Clinical follow-up may be obtained at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual cared for in the UC Davis Health System
* disorders of lipoproteins or arteriosclerosis

Exclusion Criteria:

* Subjects will be excluded only if they refuse to be in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will mainly include individuals who are scheduled to undergo cardiac catheterization at UC Davis Medical Center, but may include other eligible individuals. Subjects may also include individuals who have objective evidence of the extent of arteriosclerosis of the coronary, femoral or carotid arteries.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rogers, MD, Principal Investigator — University of California, Davis

REFERENCES:
- See also: UCDavis Health System — http://www.ucdmc.ucdavis.edu/clinicaltrials